CLINICAL TRIAL: NCT01678417
Title: A Phase II Study of 131I-rituximab for Patients With Relapsed or Refractory Follicular or Mantle Cell Lymphoma
Brief Title: 131I-rituximab for Relapsed or Refractory Follicular or Mantle Cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korea Cancer Center Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FL or MCL 131I-rituximab RIT
Record Dates: First submitted 2012-08-30; First posted 2012-09-05 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-08

CONDITIONS: Relapsed or Refractory Follicular Lymphoma or Mantle Cell Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, Follicular; Lymphoma, Mantle-Cell | interventions — 131I-rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 131I-rituximab (Experimental): 131I-rituximab treatment interval at least 4 weeks up to maximum 6 cycles
  Interventions: Drug: 131I-rituximab

INTERVENTIONS:
Drug: 131I-rituximab

SUMMARY:
Follicular lymphoma (FL) and mantle cell lymphoma (MCL) are rare lymphomas which consist of less than 5% of non-Hodgkin lymphoma in Korea. Although FL with histologic grade 1 or 2 has relatively good prognosis, continual treatment is needed due to frequent relapse. FL with histologic grade 3 has poor prognosis similar to that of diffuse large B cell lymphoma. Meanwhile, the response rate to systemic chemotherapy in MCL is low, so the treatment of relapsed MCL is challenging. So we investigate the efficacy of radioimmunotherapy using 131I-rituximab in refractory or relapsed patients with FL or MCL

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed follicular lymphoma or mantle cell lymphoma
* relapsed or refractory patients
* Eastern Cooperative Oncology Group performance status ≤ 2
* age≥ 20 years
* More than one measurable lesion (More than 2cm sized lesion in conventional CT scan,More than 1cm sized lesion in spiral CT or contrast-enhanced PET/CT)
* Adequate renal function (serum creatinine ≤ 2.0 mg/dl or Ccr ≥ 60 ml/min)
* Adequate hepatic function (serum bilirubin ≤ 2.0 mg/dl , AST/ALT ≤ 3 upper normal limit)
* Adequate bone marrow reservoir (ANC ≥1,500/㎕, platelet count≥ 75,000/㎕)
* patient who agree the purpose and intention of this clinical trial

Exclusion Criteria:

* recent (<5 years) history of other malignancy or unrecovered from the disease (appropriately treated skin cancer and uterine cervix carcinoma in situ are excluded)
* hemodynamically unstable due to the recent (<12 months) history of severe
* heart disease such as myocardial infarction
* acute complications of severe lung or metabolic disease
* Combined severe neurological or psychiatric disease
* Unrecovered from infection or other medical disease
* Recent (<30 days) history of enrollment of other clinical trial
* Pregnant or breast-feeding woman
* women of childbearing potential and men not employing adequate contraception at least for 1 year
* previous history drug allergy to the content of 131I-rituximab
* Infection(sepsis, pneumonia, viral infection, etc) (inactivated hepatitis B carrier can be enrolled)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2012-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | up to 5 years

SECONDARY OUTCOMES:
Response duration | up to 5 years
Overall survival | up to 5 years
Number of Adverse Events | up to 5 years
progression free survival | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Hye Jin Kang, M.D., Principal Investigator — Korea Cancer Center Hospital, Korea Institute of Radiological and Medical Sciences
Locations (1):
- Korea Cancer Center Hospital, Korea Institute of Radiological and Medical Sciences, Seoul, South Korea